CLINICAL TRIAL: NCT05309915
Title: A Phase 1, Single-Center, Randomized, Dose-Escalation, Sequential Cohort Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Ascending Dose of STP707 Administered Intravenously in Healthy Subjects
Brief Title: A Study of STP707 Administered by IV in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-707-002
Record Dates: First submitted 2022-03-10; First posted 2022-04-04 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Initially, for each cohort subjects will be randomized 1:1 to STP707 or placebo. After safety evaluation up to 8 additional subjects will be enrolled randomized 7:1 to STP707 or placebo within the same cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Other): Dose 3mg of STP707 (8 subjects) + placebo (2 subjects) randomized
  Interventions: Drug: STP707
- Cohort 2 (Other): Dose 6mg of STP707 (8 subjects) + placebo (2 subjects) randomized
  Interventions: Drug: STP707
- Cohort 3 (Other): Dose 12mg of STP707 (8 subjects) + placebo (2 subjects) randomized
  Interventions: Drug: STP707
- Cohort 4 (Other): Dose 24mg of STP707 (8 subjects) + placebo (2 subjects) randomized
  Interventions: Drug: STP707

INTERVENTIONS:
Drug: STP707 — STP707 Powder for Injection, contains 2 (siRNA) and (HKP+H) delivery system.

SUMMARY:
Single center study, randomized, to evaluate safety, tolerability, PK of single ascending dose of STP707 when administered by IV infusion in healthy subjects.

DETAILED DESCRIPTION:
The study includes a screening period, admission, treatment period and follow up period.

Four doses will be evaluated in 4 cohorts with up to 10 subjects per cohort. Each individual will receive a single dose of STP707 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 55 years of age, inclusive, at the time of signing the informed consent form (ICF).
2. Subjects must be in generally reasonable health with clinically insignificant screening and admission results (medical history, 12-lead electrocardiogram [ECG], physical examination, and laboratory tests), as determined by the Investigator.
3. Subjects must have a body mass index (BMI) >18 kg/m2 or <32 kg/m2
4. Subjects must have aspartate transaminase (AST), alanine transaminase (ALT), total bilirubin (TBIL), alkaline phosphatase (ALP), and glucose within upper limit of normal (ULN) range per reference laboratory reference ranges at Screening and Day -1 (Admission); one repeat laboratory analysis allowed per Investigator discretion.
5. Women of childbearing potential must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 (Admission), must not be actively breastfeeding, or planning to become pregnant during the study, and if not practicing abstinence from heterosexual activity that could result in conception (if this is the preferred and usual lifestyle of the subject), must agree to use 2 approved methods of birth control, during the study and for at least 60 days after the last dose of study drug, from the list below:

   1. Condom plus diaphragm.
   2. Condom plus cervical cap or female condom.
   3. Hormonal contraceptives (stable dose for 28 days [4 weeks] prior to Screening) plus condom.
   4. Intrauterine device (in place for 28 days [4 weeks] prior to Screening) plus condom.
   5. Condom plus spermicide.
   6. Partner vasectomy and use of barrier contraception methods (e.g., male condom, diaphragm, or sponge with spermicide).
6. Women of nonchildbearing potential must be either surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/salpingectomy) or >1 year postmenopausal with follicle-stimulating hormone (FSH) in the postmenopausal range and not actively breastfeeding.
7. Men must agree to use barrier contraception (condom with spermicide) and refrain from sperm donation from the first dose of study drug until at least 90 days after the last dose of study drug. Post vasectomy, men must agree to use a barrier method (or partner barrier method) from the first dose of study drug until at least 90 days after the last dose of study drug.
8. Subjects must be informed of the nature of the study and must have agreed to and be able to read, review, and sign the study ICF prior to any study related procedure being performed.

Exclusion Criteria:

1. Current or previous cancer, excluding basal cell carcinoma that has been in remission for >5 years prior to dosing and in situ cervical carcinoma; diabetes or known diagnosis of prediabetes; or any clinically significant cardiovascular (including ECG disturbances or history of rhythm disturbance/abnormality), endocrine, renal, hepatic, gastrointestinal, hematologic, respiratory, dermatological, neurological, psychiatric, or other disorder.
2. Hypertension, defined as blood pressure >140/90 mmHg (2 separate readings at least 15 minutes apart if first reading is not within normal range).

   a. NOTE: For the Screening blood pressure measurement, subjects should avoid smoking, caffeine, or exercise within 30 minutes prior to measurement; empty his or her bladder; then sit quietly in a comfortable chair with back support for at least 5 minutes prior to blood pressure measurement; and remain still during the measurement. Blood pressure should be measured with the subject's limb supported, with the blood pressure cuff at heart level, and with the correct cuff size. The measurement should not be taken over clothes.
3. Hyperlipidemia defined as

   1. Cholesterol >300 mg/dL.
   2. Low-density lipoprotein cholesterol >190 mg/dL.
   3. And/or triglycerides >500 mg/dL. Note: Abnormal laboratory values may be repeated once at Investigator discretion.
4. Hemoglobin A1c (HbA1c) >6.5% at Screening. Note: Abnormal laboratory values may be repeated once at Investigator discretion.
5. Hemoglobin or hematocrit outside upper and lower limits of normal range per reference laboratory range at both Screening and Day -1 (Admission).
6. Creatinine kinase (CK) > ULN at Screening and Day-1 (Admission).
7. Serum creatinine above upper limit of normal range per reference laboratory reference ranges at both Screening and Day -1 (Admission). Note: Abnormal laboratory values may be repeated once at Investigator discretion.
8. Estimated glomerular filtration rate < 90 mL/min/1.73 m2 (calculated using the Chronic Kidney Disease Epidemiology Collaboration equation) at Screening and Day-1 (Admission). One retest of the exclusionary eGFR value is allowed at the discretion of the Investigator.
9. Known sensitivity or allergies to Trehalose; history of severe hypersensitivity to IV infusion.
10. Unwillingness to abstain from alcohol for 72 hours prior to dosing through EOS/ET.
11. Use of prescription or nonprescription drugs (excluding hormonal contraceptives), if clinically applicable, including vitamins, supplements, herbal preparations, and medicines that prolong QT/QTc within 7 days or 5 times longer than the half-life (whichever is longer) prior to the first dose of study drug through EOS (approximately 60 days).
12. Blood or plasma donation within 60 days prior to dosing.
13. Use of live and non-live vaccine within 30 days prior to the first dose of study drug or an intention to receive such a vaccine at any time during the study.
14. Received an investigational agent in another clinical study within 30 days prior to the first dose of study drug, or within 10 times longer than the half-life of the compound with which the subject was treated, whichever is longer.
15. Positive results of any of the virology tests (human immunodeficiency virus (HIV test), hepatitis B virus (HBsAg test) or hepatitis C virus (hepatitis C antibody test).
16. Diagnosed to be COVID-19 positive by polymerase chain reaction testing (SARS CoV 2 RT PCR positive) of a respiratory specimen (preferably a nasopharyngeal swab) on Day -2.

    NOTE: Rapid Antigen Test may be used if PCR testing is unavailable
17. Personal or family history of vascular aneurysms and disorders.
18. Personal or family history of long QT syndrome.
19. Personal or family history of hypokalemia.
20. Corrected QT interval using Fridericia's formula (> 450 msec) based on the average of triplicate ECGs.
21. History of alcoholism or abuse within 2 years prior to Screening.
22. Positive urine drug or breath alcohol screen at Screening or Day -1 (Admission).
23. Any condition that, in the opinion of the Investigator, would complicate or compromise the study data or the well-being of the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluate safety & tolerability of STP707 when administered by IV in healthy subjects | 60 DAys
  Number and percentage of subjects in total experiencing treatment-emergent (AEs) from baseline.
Evaluate safety & tolerability of STP707 when administered by IV in healthy subjects | 60 days
  Number and percentage of subjects in each dose cohort experiencing treatment-emergent (AEs) from baseline.

SECONDARY OUTCOMES:
Evaluate (PK) of STP707 when administered by IV in healthy subjects | 60 Days
  PK parameters will be computed from individual plasma concentrations of STP707. Plasma concentrations will be assessed at each time point by study visit and cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lebel, MD, Study Director — Chief Medical Officer
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No